CLINICAL TRIAL: NCT00095472
Title: Therapeutic Application of Intravascular Nitrite for Sickle Cell Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 050016; 05-H-0016
Record Dates: First submitted 2004-11-04; First posted 2004-11-05 (Estimated); Last update posted 2019-11-05 (Actual); Status verified 2015-12-07

CONDITIONS: Sickle Cell Anemia
Keywords: Blood Flow; Nitric Oxide; Vascular Function; Vasodilation; Vaso-Occlusive Pain Crisis; Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell; Aneurysm | interventions — omega-N-Methylarginine; Sodium Nitrite

INTERVENTIONS:
Drug: L-NMMA
Drug: Sodium Nitrite

SUMMARY:
This study examines ways in which nitric oxide (NO), an important molecule that controls how blood flows through the body's vessels, might be restored with a compound called sodium nitrite. It is hoped that the result will reverse the effect of decreased flow of blood due to sickled cells-that is, cells that have changed into the shape of a crescent or sickle. Sickle cell disease is the most common genetic disease affecting African Americans. About 8% of that population has the sickle cell trait. The changed cells can become attached to blood vessels, decreasing blood flow to vital organs. There can be the loss of needed proteins, including hemoglobin, that deliver oxygen throughout the body.

Adults at least 18 years of age who have the SS form of sickle cell disease or S-beta-thalassemia, are in either a steady state or crisis, give informed and written consent for participation, and have had a negative pregnancy test may be eligible for this study. Adults with any other disease that puts them at risk for reduced circulation are not eligible. Women who are breastfeeding are not eligible.

Participants will undergo a medical history, including family medical history, and a detailed physical evaluation, to take about 1 hour. There will be a collection of blood; echocardiogram, which involves taking a picture of the heart and its four chambers; and measurement of exhaled carbon monoxide, carbon dioxide, and NO. A procedure called orthogonal polarization spectral imaging will be performed. A small object the size of a Popsicle stick will be placed under the tongue or on a fingertip. This procedure presents a picture of blood flow and how the red blood cells appear as they circulate through blood vessels. The study will be conducted in the Vascular Laboratory/Cardiovascular Floor or Intensive Care and will last about 4 hours.

During the study, patients will lie in an adjustable reclining bed and chair. Small tubes will be placed in the artery and vein of the forearm at the inside of the elbow. A small pressure cuff will be applied to the wrist and a larger one to the upper arm. Both cuffs will be inflated with air. A strain gauge, resembling a rubber band, will go around the widest part of the forearm. When the pressure cuffs fill with air, blood will flow into the arm, and information from the strain gauge will be recorded. Between administrations of each medicine, there will be 30-minute rests. Normal saline will be put into the small tube in the artery. Measurements of the blood flow in the forearm will be taken, and a small blood sample will be taken to measure blood counts, proteins, and other natural body chemicals. Then a medicine called sodium nitroprusside, which causes blood vessels to expand and increase blood flow, will be placed into the forearm. It will be given at three different doses for 3 minutes each, with measurements recorded after each dose. Then a medicine called L-NMMA will be placed into the forearm. L-NMMA generally decreases local blood flow by preventing nitric oxide from being produced in the cells lining the blood vessels. It will be given at two different doses for 5 minutes each, with blood flow measured after each dose. Next, nitrite will be placed in the forearm at three different doses for 5 minutes each. Before and after nitrite is given, the researchers will measure the amount of the NO, carbon monoxide, and carbon dioxide that the patients breathe out. Then the procedure for administering normal saline, sodium nitroprusside, and L-NMMA will be repeated, as will a blood test.

This study will not have a direct benefit for participants. However, it is hoped that the information gained from the study will help to develop treatment options for patients with sickle cell disease.

DETAILED DESCRIPTION:
Sickle cell disease is an autosomal recessive disorder and the most common genetic disease affecting African-Americans. Approximately 0.15% of African-Americans are homozygous for sickle cell disease, and 8% have sickle cell trait. Hemoglobin S polymerization leads to red cell rigidity, microvascular obstruction, inflammation, and end-organ ischemia-reperfusion injury and infarction. Our published data indicate that up to 50% of sickle cell patients have endothelial dysfunction due to impaired bioavailability of endogenous nitric oxide due in large part to scavenging of nitric oxide by cell-free plasma hemoglobin. These data suggest that therapies directed at restoring NO bioavailability might prove beneficial. We have recently discovered that the nitrite anion, available currently for human use as a component of the cyanide antidote kit, is a vasodilator in vivo by generating nitric oxide (NO) in tissues with lower oxygen tension and pH. The mechanism involves a novel physiological function of human hemoglobin as an oxygen- and pH dependent nitrite reductase. To date we have observed that nitrite infusions in animal models significantly reduce liver and cardiac ischemia-reperfusion injury and infarction in mouse models, prevent cerebral vasospasm after subarachnoid hemorrhage in primates, and decrease pulmonary hypertension in newborn hypoxic sheep. The current protocol is designed as a phase I/II trial to address the hypothesis that nitrite infusions will vasodilate the circulation in patients with sickle cell disease at rest and during vaso-occlusive pain crisis, inactivate circulating cell-free plasma hemoglobin, reduce pulmonary artery pressures and reduce ischemia-reperfusion injury (measured by circulating markers of oxidant stress).

ELIGIBILITY:
* INCLUSION CRITERIA:

Must be at least 18 years of age

Homozygous sickle cell disease or S beta-0-thalassemia/alpha-thalassemia

Provides informed, written consent for participation

EXCLUSION CRITERIA:

Patients with currently uncontrolled hypertension (diastolic blood pressures greater than 95 mmHg)

Hypercholesterolemia (LDL cholesterol greater than 130 mg/dL)

Diabetes mellitus (fasting blood glucose greater than 120 mg/dL)

Smoking within one month

Dietary ingestions of herbal medications, alcohol or caffeine within 12 hours of the study

Arteriosclerotic cardiovascular disease

Peripheral arteriosclerotic vascular disease

Treatment within the last 14 days with sildenafil, vardenafil, tadalafil, inhaled nitric oxide, nitroglycerin or other NO-dependent drugs, such as arginine

Red cell G6PD activity below normal range (All subjects will be tested for red blood cell G6PD deficiency; levels below the lower limits of normal will result in exclusion from participation in the study)

Cytochrome B5 deficiency

History of reaction to a medication or other substance characterized by dyspnea and cyanosis

Lactating females (Lactating females will not participate since nitrites cross into breast milk and could cause methemoglobinemia in the infant)

Pregnancy testing (urine or blood) will be required of all women of reproductive age to exclude current pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2004-11-01; Primary Completion 2007-08-24 (Actual); Study Completion 2007-08-24 (Actual)

PRIMARY OUTCOMES:
Determine the potential therapeutic effect of intra-arterial nitrite infusion to restore nitric oxide dependent regional blood flow in patients with sickle cell disease.

CONTACTS AND LOCATIONS:
Overall Officials: John F Tisdale, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Furchgott RF, Zawadzki JV. The obligatory role of endothelial cells in the relaxation of arterial smooth muscle by acetylcholine. Nature. 1980 Nov 27;288(5789):373-6. doi: 10.1038/288373a0. PMID 6253831
- [Background] Ignarro LJ, Byrns RE, Buga GM, Wood KS. Endothelium-derived relaxing factor from pulmonary artery and vein possesses pharmacologic and chemical properties identical to those of nitric oxide radical. Circ Res. 1987 Dec;61(6):866-79. doi: 10.1161/01.res.61.6.866. PMID 2890446
- [Background] Rees DD, Palmer RM, Hodson HF, Moncada S. A specific inhibitor of nitric oxide formation from L-arginine attenuates endothelium-dependent relaxation. Br J Pharmacol. 1989 Feb;96(2):418-24. doi: 10.1111/j.1476-5381.1989.tb11833.x. PMID 2924084